CLINICAL TRIAL: NCT07030881
Title: Effect of Spacer Use on Exacerbation Risk in High-Risk Older Adults With Chronic Airway Diseases Receiving Triple Therapy: A Multicenter Randomized Controlled Trial
Brief Title: Effect of Spacer Use on Exacerbation Risk in High-Risk Older Adults With Chronic Airway Diseases Receiving Triple Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Caochao, Principal Investigator, First Affiliated Hospital of Ningbo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-146A-01
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Asthma, COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy Group (Active Comparator): Participants will receive standard triple inhaled therapy using a pressurized metered-dose inhaler (ICS/LABA/LAMA). They will receive routine inhalation technique training but will not use a spacer device.
  Interventions: Drug: pMDI Triple Inhaler Only
- Spacer Group (Experimental): Participants will receive the same standard triple inhaled therapy via pMDI (ICS/LABA/LAMA) plus a valved mouthpiece spacer. Inhalation technique training will include proper spacer usage, including attachment, mouth seal, actuation timing, and cleaning. The spacer is intended to optimize pulmonary drug delivery, reduce the need for hand-breath coordination, and minimize local side effects.
  Interventions: Drug: pMDI Triple Inhaler and Spacer

INTERVENTIONS:
Drug: pMDI Triple Inhaler and Spacer — Participants in this group will use a valved mouthpiece spacer in combination with standard triple inhaled therapy delivered by a pressurized metered-dose inhaler (ICS/LABA/LAMA). The spacer device helps reduce the need for hand-breath coordination, prolongs aerosol suspension time, and improves drug delivery to the lungs. Participants will be trained in proper spacer use, including device attachment, timing of actuation and inhalation, mouth seal technique, cleaning, and daily maintenance. This intervention aims to optimize inhalation technique, improve treatment adherence, and potentially reduce the incidence of moderate-to-severe exacerbations.
  Arms: Spacer Group
Drug: pMDI Triple Inhaler Only — Participants in the control group will receive a standard fixed-dose combination of inhaled corticosteroid (ICS), long-acting beta-agonist (LABA), and long-acting muscarinic antagonist (LAMA) administered via pressurized metered-dose inhaler (pMDI). No spacer will be used. All participants will receive standardized inhalation technique training at baseline, including hand-held device usage, actuation-inhalation timing, breath-hold, and mouth rinsing. This group represents the current standard-of-care for stable, high-risk COPD or asthma patients as per GOLD and GINA guidelines.
  Arms: Standard Therapy Group

SUMMARY:
This study evaluates whether adding a spacer device to triple inhaled therapy (ICS/LABA/LAMA via pMDI) can reduce acute exacerbations in elderly patients (≥65 years) with stable chronic airway diseases (COPD or asthma) who are classified as high-risk based on GOLD or GINA guidelines. High-risk is defined as ≥1 hospitalization or ≥2 moderate exacerbations in the past 12 months.

Despite receiving maximum inhaled treatment, these patients often have poor inhaler technique due to age-related limitations. A spacer may improve drug delivery, adherence, and reduce local side effects.

In this multicenter, open-label, randomized controlled trial, 380 participants will be assigned to standard therapy with or without a valved face-mask spacer. The primary outcome is the 3-month incidence of moderate-to-severe exacerbations. Secondary outcomes include lung function, adherence, inhalation technique, side effects, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years, no gender restriction;
2. Confirmed diagnosis of chronic obstructive pulmonary disease (COPD) based on GOLD criteria or bronchial asthma based on GINA criteria;
3. Currently on stable treatment with fixed-dose combination ICS/LABA/LAMA via pMDI for ≥4 weeks;
4. History of any of the following in the past 12 months:

   1. ≥1 hospitalization due to exacerbation, or
   2. ≥2 moderate exacerbations requiring systemic corticosteroids and/or antibiotics;
5. Able to complete inhalation technique training and demonstrate basic communication and device-handling abilities;
6. Provides written informed consent to participate in the study.

Exclusion Criteria:

1. Use of other inhalation devices as primary therapy (e.g., DPI, SMI, or nebulizer);
2. Regular use of a spacer device for ≥3 weeks within 3 months prior to enrollment;
3. Current or recent (within 4 weeks) acute exacerbation not fully resolved;
4. Severe cognitive impairment (MMSE score <18);
5. Presence of severe systemic comorbidities (e.g., end-stage malignancy, advanced heart failure, hepatic or renal failure);
6. Participation in another interventional clinical trial;
7. Inability to use a mouthpiece-based spacer (e.g., structural oral/facial abnormalities, severe anxiety);
8. Known allergy or hypersensitivity to spacer device materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Moderate-to-Severe Acute Exacerbations Within 3 Months | Baseline, 3 months
  Moderate exacerbation is defined as a worsening of respiratory symptoms requiring treatment with systemic corticosteroids and/or antibiotics. Severe exacerbation is defined as requiring emergency department visit or hospitalization. All events must be confirmed by the treating physician and recorded in the case report form (CRF). This outcome evaluates whether the use of a valved spacer reduces the rate of such events compared to standard therapy alone.

SECONDARY OUTCOMES:
Change in Post-Bronchodilator FEV₁ From Baseline to 3 Months | Baseline and 3 months
  FEV₁ (forced expiratory volume in 1 second) will be measured using a standardized spirometer following ATS/ERS guidelines. Change will be assessed as both absolute value and percentage improvement. A clinically meaningful improvement is defined as an increase of ≥100 mL or ≥12% from baseline.
Change in Treatment Adherence Score (MARS-5) From Baseline to 3 and 6 Months | Baseline, 3 months, and 6 months
  The Medication Adherence Report Scale (MARS-5), a validated 5-item questionnaire (score range: 5-25), will be used to assess adherence. Improvement is defined as an increase of ≥3 points from baseline.
Time to First Moderate-to-Severe Acute Exacerbation | Baseline, 3 months
  Time from randomization to first moderate or severe exacerbation will be recorded. Kaplan-Meier survival analysis will be used to compare groups. Events will be defined per GOLD/GINA criteria and confirmed by treating physicians.
Change in Inhalation Technique Score From Baseline to 3 Months | Baseline, 3 months
  Inhalation technique will be scored using a structured checklist (5 items × 5 points, total score 25). Components include device handling, breath-hold, actuation timing and cleaning. Improvement is defined as an increase of ≥5 points.
Change in Local Side Effect Score (ICS-Related) | Baseline, 1, 2, 3 months
  Monthly assessments of local side effects related to ICS will be recorded, including throat irritation, hoarseness, and oral discomfort. Each symptom will be rated on a 0-10 scale (0 = none, 10 = severe).
Change in Patient Satisfaction Score (VAS) | 3 and 6 months
  A visual analog scale (VAS, range 0-10) will be used to assess satisfaction with the inhalation treatment method. Higher scores indicate greater satisfaction.
Asthma Control Level Based on Four GINA-Recommended Indicators | Baseline and 3 months
  For asthma patients, control status will be evaluated based on four criteria: daytime symptoms >2/week, nighttime awakening, reliever use >2/week, and activity limitation. Control will be categorized as: well-controlled (0), partly controlled (1-2), or uncontrolled (≥3).

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Anhui Chest Hospital, Hefei
  - Beilun District Second People's Hospital, Ningbo
  - Fenghua District People's Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Xiangshan First People's Hospital Medical and Health Group, Ningbo
  - Ninghai County First Hospital, Ninghai
  - Taizhou Municipal Hospital, Taizhou

IPD SHARING:
Plan to Share IPD: No